CLINICAL TRIAL: NCT01070225
Title: Reversal of Acute β-Blocker Induced Bronchoconstriction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHO001
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Hydrocortisone; Propranolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone and Propranolol (Experimental): Participant administered 10 or 20mg propranolol orally. Participants meeting the parameters are randomised to receive 400mg Hydrocortisone intravenously. Participant then receives Histamine PC10 challenge, Administered 5mg Salbutamol via nebuliser, administered 500mcg Ipratropium Bromide via nebuliser; visit end
  Interventions: Drug: Hydrocortisone/ Placebo and Propranolol
- Placebo and propranolol (Placebo Comparator): identical to other arm but participant receive placebo injection as opposed to hydrocortisone
  Interventions: Drug: Hydrocortisone/ Placebo and Propranolol

INTERVENTIONS:
Drug: Hydrocortisone/ Placebo and Propranolol — Hydrocortisone 400mcg Propranolol 10mg or 20 mg

SUMMARY:
Current therapies for the management of asthma include inhalers. Types of these medications (beta agonists), improve asthma symptoms by stimulating areas (receptors) within the human airway resulting in dilation of the human airway. Whilst these drugs are highly effectively in the immediate setting their longterm use, constantly stimulation of receptors within the airway has been associated with increased asthma exacerbations and rare cases of death.

Conversely medications that block receptors within the human airway (betablockers)have been avoided in asthma.

The main reason for this is because of the possible acute airway narrowing that can occur after soon after administration. However chronic use of betablockers in asthma has recently been shown to be of benefit in reducing airway inflammation which is of great importance in improving asthma control and reducing symptoms.

Despite this early evidence supporting chronic use of beta blockers in asthma, there is concern in 2 major regards:their potential to cause acute airway narrowing (irrespective of longterm benefit) and the possibility that they could block the reliever action of beta agonists.

The objective of this study is to establish how best to reverse the short term effects of a single dose of beta blocker.

This study is designed as a single centre study, with participants attending the department on approximately 3 separate visits (including a screening visit) at approximately 1 weekly intervals.

DETAILED DESCRIPTION:
Asthma was originally thought to be associated with an intrinsic defect of β2- adrenoceptor function tipping the balance towards parasympathetic bronchoconstriction. While β2-agonists are highly effective for the acute relief of bronchoconstriction, their chronic use is accompanied by an adaptive reduction in β2ADR numbers and associated desensitisation of response, resulting in increased exacerbations and rare cases of death. Conversely the chronic use of β blockers have been shown in murine models to reduce airway inflammation and mucous metaplasia. Recent work in humans has further demonstrated a potential benefit of β blockers in asthmatics by demonstrating a significant improvement in airway hyperresponsiveness to bronchial challenge1.

Despite this early evidence supporting chronic use of β blockers in asthma, there is concern in 2 major regards: their potential to cause acute bronchoconstriction (irrespective of long-term benefit) and the possibility that they could block the reliever action of β-agonists.

Sub-sensitivity of β-adrenoceptors occurs following treatment with long-acting β-agonists. Previous work in our department has shown that high dose steroids can re-establish the β-adrenoceptor function following such down-regulation2. It therefore seems plausible that a similar response may occur following β-blockade (reversing β-blockade and re-establishing β-agonist sensitivity).

The investigators wish to gather evidence for the best methods to treat β-blocked patients in the short term. The investigators therefore wish to examine the effects of acute-β blockade with low dose propranolol on mild-to-moderate asthmatics. The investigators wish to simulate airway stress and rescue in acutely β-blocked patients. For safety purposes the investigators have chosen propranolol due to its short half-life of 3 to 5 hours. Importantly the ability to achieve airway reversibility and recovery following acute β-blockade will influence the long term viability of chronic β blockers use in the management of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to obtain Informed consent.
* Mild to Moderate Asthmatics taking ≤1000μg BDP per day or equivalent.
* Histamine PC10
* Ability to perform spirometry, IOS, bronchial challenge and all domiciliary measurements.
* Withhold LABAs, montelukast and theophyllines for 1 week prior to study.
* FEV1 >80% predicted with diurnal FEV1 variation <20% post wash out.

Exclusion Criteria:

* Uncontrolled symptoms of asthma.
* Resting BP<110 systolic or HR<60.
* Pregnancy or lactation.
* Known or suspected sensitivity to IMP.
* Inability to comply with protocol.
* Any degree of heart block.
* Rate limiting medication including β blockers, rate limiting Calcium Channel Blockers and Amiodarone.
* Any other clinically significant medical condition that may either endanger the health or safety of the participant, or jeopardise the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To establish whether acute β-blockade influences the ability to achieve airway reversibility and recovery with systemic corticosteroids and nebulised bronchodilators following histamine challenge in mild to moderate asthmatics. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Lipworth, MD, Principal Investigator — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, Unviersity of Dundee, Dundee, United Kingdom

REFERENCES:
- [Result] Short PM, Williamson PA, Lipworth BJ. Effects of hydrocortisone on acute beta-adrenoceptor blocker and histamine induced bronchoconstriction. Br J Clin Pharmacol. 2012 May;73(5):717-26. doi: 10.1111/j.1365-2125.2011.04143.x. PMID 22077869